CLINICAL TRIAL: NCT05948605
Title: Evaluation of the Empower Neuromodulation System for the Treatment of Alcohol Use Disorder
Brief Title: EMPOWER AUD Pivotal Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRD-12-1477-01
Record Dates: First submitted 2023-05-12; First posted 2023-07-17 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alcoholism; Alcohol Abuse; Alcohol Use Disorder
Keywords: Alcoholism; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Multi-center, double-blinded, prospective, randomized, sham-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Site staff are blinded to the subject's assigned Arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Treatment (Active Comparator): The Active Treatment will use a functional Stimulator system.
  Interventions: Device: Empower Neuromodulation System
- Sham Treatment (Sham Comparator): The Sham Treatment (Placebo) will use a functional Stimulator system, but will provide a treatment in a location that is believed to have no benefit or harm to the subject.
  Interventions: Device: Empower Neuromodulation System

INTERVENTIONS:
Device: Empower Neuromodulation System — The Empower Neuromodulation System is designed to provide transcutaneous stimulation to the branches of a spinal nerve. The system comprised of three key components: (A) The Stimulator, (B) the Empower smartphone app, and (C) the Gel Patch. The smartphone application is used to coordinate treatment and record participant responses.

SUMMARY:
Multi-site, double-blinded, prospective, randomized, sham-controlled study

DETAILED DESCRIPTION:
To evaluate the safety and effectiveness of the Empower Neuromodulation System in alcohol use disorder (AUD) patients. The primary safety endpoint will be device-related serious adverse events. The primary effectiveness endpoint will be responder rate at 12 weeks, where a responder is defined as a subject who experiences at least a one level reduction in the WHO risk level for daily alcohol consumption from Baseline to Week 12 as measured via the 28-day Timeline Follow-back (TLFB). Responder rate will be compared between subjects randomized to the active treatment vs. the sham treatment.

ELIGIBILITY:
Inclusion Criteria:

A candidate for this study must meet ALL of the following inclusion criteria:

* Women and men ≥21 years of age
* Individual has a current diagnosis of alcohol use disorder per DSM-5 via M.I.N.I. assessment by clinician
* Individual has a desire to reduce or quit alcohol use
* Based on the 28-day TLFB at enrollment, individual has an average daily alcohol consumption in the WHO risk levels of moderate, high, or very high (men: ≥2.91 drinks/day; women: ≥1.41 drinks/day)
* Individual has a breath alcohol concentration of 0.02% or less at enrollment
* Individual has a negative urine pregnancy test at screening (females of childbearing age only)
* Individual is able to provide informed consent
* Individual is capable and willing to follow all study-related procedures

Exclusion Criteria:

A candidate will be excluded from the study if ANY of the following conditions are met:

* Individual has a current, unstable psychiatric disorder per DSM-5 via M.I.N.I. assessment that is clinically significant enough to preclude study participation per the judgment of the study site PIs
* Individual has been diagnosed with a neurodegenerative disease, including Parkinson's disease, dementia, and Alzheimer's disease
* Individual has a current substance use disorder (SUD) diagnosis other than alcohol, nicotine, or cannabis per DSM-5 via M.I.N.I. assessment by clinician
* Individual requires acute medical detoxification from alcohol per based on a score of 12 or more on the Clinical Institute Withdrawal Assessment Alcohol Scale Revised (CIWA-Ar)
* Individual is taking or plans to start taking an AUD pharmacotherapy during the study
* Individual has had a change in AUD pharmacotherapy in the past 4 weeks
* Individual has initiated or discontinued SUD psychotherapy in the past 4 weeks, has had a change in SUD psychotherapy modality in the past 4 weeks, or expects to initiate, discontinue, or change psychotherapy modality during the study
* Individual has an active implant and/or an implanted electrical or neurostimulator device (e.g., pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, sacral stimulator, bone growth stimulator, or cochlear implant)
* Individual is currently using, or has used in the past 3 months, transcutaneous electrical nerve stimulation (TENS) in the upper extremities
* Individual is currently receiving, or has received in the past 3 months, acupuncture, or acupressure in the upper extremities
* Individual has an electrically conductive metal object (e.g., jewelry) that cannot be removed and will directly contact the gel electrodes of the Empower Neuromodulation System at either treatment location
* Individual has an open incision, wound, scar, active infection or otherwise compromised skin at the treatment locations and will directly contact the gel electrodes of the Empower Neuromodulation System at either anatomic location
* Individual has a history of epilepsy or a seizure disorder
* Individual has been clinically diagnosed with peripheral nerve damage of the upper limbs or has numbness or tingling in an upper limb at least weekly
* Individual is female and currently pregnant or breastfeeding, has been pregnant within the past 6 months, intends to become pregnant during participation in the study, or is unwilling to practice birth control during participation in the study
* Individual will not, for the duration of participation in the study, have a living situation that provides regular access to an electrical outlet for charging the study device and smartphone
* Individual has used an investigational drug, biologic, or medical device in the past 4 weeks
* Individual is deemed unsuitable for enrollment in the study by the investigator based on the subject's history or physical examination

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Frequency of device-related Serious AEs (SAEs) | Week 12
  The primary safety endpoint will be comparing the frequency of device-related Serious AEs (SAEs) between the Active and Sham Treatment groups, where device-related SAEs include probably and possibly device-related serious adverse events
Primary Effectiveness Endpoint: Change in WHO risk level via 28-day TLFB | Week 12
  The primary effectiveness endpoint is the responder rate at Week 12, where a responder is a study subject who experiences ≥1 level reduction in the WHO risk level from Baseline to Week 12 via the 28-day Timeline Follow-back (TLFB), and responder rate is the percentage of participants in a treatment group who are responders

SECONDARY OUTCOMES:
Change in Alcohol Craving Intensity via the Penn Alcohol Craving Survey (PACS) | Week 12
  Change in alcohol craving intensity. The change in alcohol craving intensity as assessed via the Penn Alcohol Craving Survey (PACS) from Baseline to Week 12 will be compared between the Active and Sham Treatment groups. The scale has a range of 0-30 where a higher score indicates more severe cravings.
Change in Heavy Drinking Days (HDD) via 28-day TLFB | Week 12
  Change in heavy drinking days (HDD). The change in HDD as assessed via the 28-day Timeline Follow-Back (TLFB) from Baseline to Week 12 will be compared between the Active and Sham Treatment groups, where a HDD is defined as 5 or more drinks for men and 4 or more drinks for women in one calendar day
Change in Alcohol Related Problems via SIP | Week 12
  Change in alcohol-related problems. The change in alcohol-related problems as assessed via the Short Index of Problems (SIP) from Baseline to Week 12 will be compared between the Active and Sham Treatment groups. The total score has a range of 0-15 where a higher total indicates more problems.
Change in Alcohol Consumption via PEth analysis | Week 12
  Change in phosphatidylethanol (PEth)-based evaluation of alcohol consumption. The change in alcohol consumption as assessed via PEth analysis from Baseline to Week 12 will be compared between the Active and Sham Treatment groups.
Change in Alcohol Craving Intensity via daily self reports | Week 12
  Change in daily alcohol craving intensity. The change in daily alcohol craving intensity as assessed via daily self-reports on the Empower app (100-point Visual Analog Scale (VAS)) from Week 1 to Week 12 will be compared between the Active and Sham Treatment groups. The scale range is 0-100, where the higher rating indicates higher level of alcohol cravings.
Improvement in Clinician Assessment of Illness via CGI | Week 12
  Improvement in clinician assessment of illness. The clinician assessment of improvement in illness as assessed via Clinical Global Impression (CGI) at Week 12 will be compared between the Active and Sham Treatment groups.

OTHER OUTCOMES:
Exploratory Effectiveness - Responder Rate Week 6 | Week 6
  Responder rate at Week 6. The percentage of responders at 6 weeks will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - Drink reduction Week 12 via TLFB | Week 12
  Change in alcoholic drinks consumed at Week 12. The change in average alcoholic drinks consumed per day as assessed via the 28-day TLFB from Baseline to Week 12 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - % Drink change Week 12 via TLFB | Week 12
  Percent reduction in alcoholic drinks consumed at Week 12. The percent change in average alcoholic drinks consumed per day as assessed via the 28-day TLFB from Baseline to Week 12 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - Drinks change at Week 6 | Week 6
  Change in alcoholic drinks consumed at Week 6. The change in average alcoholic drinks consumed per day as assessed via the 28-day TLFB from Baseline to Week 6 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - Drink change Week 12 via App | Week 12
  Change in alcoholic drinks consumed at Week 12. The change in average alcoholic drinks consumed per day as assessed via the daily self-reports on the Empower app from Baseline to Week 12 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - % Drink change Week 12 via App | Week 12
  Percent change in alcoholic drinks consumed at Week 12. The percent change in average alcoholic drinks consumed per day as assessed via the daily self-reports on the Empower app from Baseline to Week 12 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - Drink change Week 6 via App | Week 6
  Change in alcoholic drinks consumed at Week 6. The change in average alcoholic drinks consumed per day as assessed via the daily self-reports on the Empower app from Baseline to Week 6 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - Change in HDD at Week 6 via TLFB | Week 6
  Change in HDD at Week 6. The change in HDD as assessed via the 28-day TLFB from Baseline to Week 6 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - Abstinence at Week 12 via TLFB | Week 12
  Abstinence at Week 12. The percent of subjects who are abstinent at Week 12 as assessed via the 28-day TLFB at Week 12 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - Alcohol consumption at Week 6 via PEth | Week 6
  Change in PEth-based evaluation of alcohol consumption at Week 6. The change in alcohol consumption as assessed via PEth analysis from Baseline to Week 6 will be compared between the Active and Sham Treatment groups.
Exploratory Effectiveness - Alcohol craving reduction at Week 6 via PACS | Week 6
  Change in alcohol craving intensity at Week 6. The change in alcohol craving intensity as assessed via the Penn Alcohol Craving Scale (PACS) from Baseline to Week 6 will be compared between the Active and Sham Treatment groups. The scale has a range of 0-30 where a higher score indicates more severe cravings.
Exploratory Effectiveness - Alcohol craving at Week 12 via PACS | Week 12
  Percent change in alcohol craving intensity at Week 12. The percent change in alcohol craving intensity as assessed via the PACS from Baseline to Week 12 will be compared between the Active and Sham Treatment groups. The scale has a range of 0-30 where a higher score indicates more severe cravings.
Exploratory Effectiveness - Alcohol craving change at Week 6 via VAS | Week 6
  Change in daily alcohol craving intensity at Week 6. The change in daily alcohol craving intensity as assessed via daily self-reports on the Empower app (100-point Visual Analog Scale (VAS)) from Week 1 to Week 6 will be compared between the Active and Sham Treatment groups. For each subject, the average craving score per day will be calculated for each study week from the daily surveys, and the average score for Week 1 will be compared against the average score for Week 6. The scale range is 0-100, where the higher rating indicates higher level of alcohol cravings.
Exploratory Effectiveness - Alcohol craving % change at Week 12 via VAS | Week 12
  Percent reduction in daily alcohol craving intensity at Week 12. The percent change in daily alcohol craving intensity as assessed via daily self-reports on the Empower app (100-point Visual Analog Scale (VAS)) from Week 1 to Week 12 will be compared between the Active and Sham Treatment groups. For each subject, the average craving score per day will be calculated for each study week from the daily surveys. The scale range is 0-100, where the higher rating indicates higher level of alcohol cravings.
Exploratory Effectiveness - Change in alcohol-related problems at Week 6 via SIP | Week 6
  Change in alcohol-related problems at Week 6. The change in alcohol-related problems as assessed via the SIP from Baseline to Week 6 will be compared between the Active and Sham Treatment groups. The total score has a range of 0-15 where a higher total indicates more problems.
Exploratory Effectiveness - Change in anxiety at Week 12 via BAI | Week 12
  Change in anxiety at Week 12. The change in anxiety as assessed via the Beck Anxiety Inventory (BAI) from Baseline to Week 12 will be compared between the Active and Sham Treatment groups. The total score has a range of 0-63 where a higher total indicates more severe anxiety.
Exploratory Effectiveness - Change in depression at Week 12 via PHQ-9 | Week 12
  Change in depression at Week 12. The change in depression as assessed via the Patient Health Questionnaire (PHQ-9) from Baseline to Week 12 will be compared between the Active and Sham Treatment groups. The questionnaire scoring ranges from 0-27 where the higher number indicates higher level of depression.
Exploratory Effectiveness - Satisfaction with treatment at Week 12 via VAS | Week 12
  Satisfaction with treatment. Satisfaction with treatment as assessed via 100-mm Visual Analog Scale (VAS) at Week 12 will be compared between the Active and Sham Treatment groups. The scale range is 0-100, where the higher rating indicates higher level of satisfaction with the device and phone app.
Exploratory Effectiveness - System Usability at Week 12 via SUS | Week 12
  Usability. System usability as assessed via the SUS at Week 12 will be compared between the Active and Sham Treatment groups. Scores from the Active Treatment group will also be compared against benchmarks for average score (SUS=68) and excellent score (SUS=80).

CONTACTS AND LOCATIONS:
Overall Officials: KT Venkateswara-Rao, PhD, Principal Investigator — TheraNova, LLC; David Pennington, PhD, Principal Investigator — Northern California Institute of Research and Education
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No